CLINICAL TRIAL: NCT02030652
Title: Impact of Synchronized Nasal Intermittent Positive Pressure Ventilation Using Non Invasive Neurally Adjusted Ventilatory Assist (NAVA) in Preterm Infants With Respiratory Distress
Brief Title: Impact of Synchronized Nasal Intermittent Positive Pressure Ventilation Using NAVA in Preterm Infants With RDS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Celso Rebello MD, MD PhD, Hospital Israelita Albert Einstein
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIAE-2013-001; 2013/12499-0 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2014-01-07; First posted 2014-01-08 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Respiratory Distress Syndrome
Keywords: premature newborn; nasal ventilation; noninvasive ventilation; continuous positive airway pressure
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SNIPPV Group (Experimental): Synchronized nasal intermittent positive pressure using NAVA ( Intermittent nasal positive pressure positive ventilation.)
  Interventions: Procedure: Intermittent nasal positive pressure positive ventilation.
- CPAP Group (Active Comparator): Nasal CPAP group without intermittent ventilation.
  Interventions: Procedure: CPAP

INTERVENTIONS:
Procedure: Intermittent nasal positive pressure positive ventilation.
  Arms: SNIPPV Group
Procedure: CPAP — Nasal continuous positive airway pressure
  Arms: CPAP Group

SUMMARY:
The nasal CPAP (continuous positive airway pressure), is a technique of noninvasive ventilation commonly used in neonatal intensive care units, and has recently been used in association with nasal intermittent mandatory ventilation (NIPPV - intermittent Nasal Positive Pressure Ventilation), which consists of the application of respiratory positive pressure cycles during the application of nasal CPAP, resulting in high pharyngeal pressures. The NIPPV has advantages over traditional CPAP, including the prevention of atelectasis, improved respiratory mechanics and decreased work of breathing in premature infants. A refinement of this technique is the use of positive pressure breaths associated with nasal CPAP synchronously in relation to the newborn's inspiratory effort (SNIPPV - Synchronized Nasal Positive Pressure Ventilation).

Synchronization allows that the cycles of inspiratory positive pressure provided by the ventilator coincide with the inspiratory effort, increasing the system efficacy. The Neurally Adjusted Ventilatory Assist (NAVA) is a mode of partial ventilatory support based on the use of electrical activity of the diaphragm (Edi) to control the mechanical ventilator. The ventilatory assistance starts according to respiratory needs of the patient, its use in very low birth weight infants showed an improvement in patient-ventilator interaction, even in the presence of leak around the endotracheal tube. This prospective randomized, clinical trial aims to evaluate, in preterm infants with gestational age lower than 34 weeks with respiratory failure treated with noninvasive ventilatory support, the impact of SNIPPV with neural adjustment (NAVA) on success ventilation and the need for endotracheal intubation when compared to treatment with traditional CPAP.

DETAILED DESCRIPTION:
Type and location of the study A prospective , randomized , open label clinical study will be conducted at the Albert Einstein Jewish Hospital Neonatal ICU, after approval by the Ethics Committee and the Research Institute of Education and Research. To participate in the study the parents or legal guardians must complete and sign the Statement of Consent.

Randomization and formation of study groups Two study groups will be formed according to the type of non- invasive ventilatory support: SNIPPV Group (synchronized nasal intermittent positive pressure) and CPAP group (continuous positive airway pressure). The formation of study groups will be by randomization through opaque envelopes containing in its interior the type of treatment to be used. The envelopes will be opened at the initiation of treatment.

Inclusion Criteria Will be included in study preterm infants with respiratory failure and indication of noninvasive ventilatory support, characterized by clinical evidence of respiratory failure requiring use of oxygen greater than or equal to a FiO2 0.25.

Exclusion Criteria Will be excluded from the study infants that parents did not agree on participation; diagnosed with major congenital anomalies; with necessity of chest drainage; diagnosis of intracranial hemorrhage grades III and IV according to the criteria of Papile et al; persistence ductus arteriosus with hemodynamic consequences and diagnosis of severe perinatal asphyxia - defined as less than 6 APGAR with 5 minutes of life.

Definition of the primary variable and secondary variables:

Demographic data regarding to birth weight, gestational age, sex, Apgar scores (1 and 5 minutes), type of delivery, use of antenatal corticosteroids, magnesium sulfate, multiple births, maternal diseases will be collected.

The main variable will be the need for endotracheal intubation. This will be defined as the need to use the fraction of inspired oxygen (FiO2) greater than 0.30 and 7 cmH2O or more of CPAP pressure for maintaining a target oxygen saturation of 88-94 % for preterm infants with gestational age less or equal to 27 6/7 weeks, or a FiO2 higher than 0.35 and 7 cmH2O or more of CPAP pressure for maintaining a target oxygen saturation of 88-94 % for preterm infants with gestational age higher or equal to 28 0/7 weeks gestation.

Secondary variables will be defined as the total time of nCPAP , the total time of oxygen use; time for the indication of invasive mechanical ventilation, the incidence of pneumothorax and the maximum values of FiO2 in noninvasive support, the average values of CPAP pressure, the incidence of bronchopulmonary dysplasia (defined as oxygen requirement at 36 weeks corrected gestational age), the incidence of intracranial hemorrhage and intracranial hemorrhage grades III and IV according to Papile et al.

Ventilatory strategies The equipment used for both ventilation modes will be the Servo i (Maquet , Getinge Group , Solna , Sweden). The pressure initially applied will be CPAP 5 cmH2O in both groups and can be increased up to 7 cm H2O at the discretion of the attending physician. The CPAP applied and FiO2 will be adjusted toward maintenance of oxygen saturation target of 88-94 % .

Statistical analysis and sample size. Comparisons between continuous variables will be performed by "t " Student test . The Kruskal - Wallys be used for non-parametric data . Categorical variables were compared using the chi -square or Fisher's exact test , as appropriate. The level of significance adopted will be 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Will be included in study preterm infants with respiratory failure and indication of noninvasive ventilatory support, characterized by clinical evidence of respiratory failure requiring use of oxygen greater than or equal to a FiO2 0.25.

Exclusion Criteria:

* Will be excluded from the study infants that parents did not agree on participation; diagnosed with major congenital anomalies; with necessity of chest drainage; diagnosis of intracranial hemorrhage grades III and IV according to the criteria of Papile et al; persistence ductus arteriosus with hemodynamic consequences and diagnosis of severe perinatal asphyxia - defined as less than 6 APGAR with 5 minutes of life.

Ages: 23 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Need for endotracheal intubation | 7 days
  Necessity of intubation and mechanical ventilation until the end of the first week of life.

SECONDARY OUTCOMES:
Total time of nCPAP | 1 month
  Total time of nCPAP use.

OTHER OUTCOMES:
Bronchopulmonary dysplasia rate | 36 weeks corrected gestational age
  Diagnosis of bronchopulmonary dysplasia

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil